CLINICAL TRIAL: NCT03910114
Title: Contrast Enhancement Characteristics of Gadolinium-Based-Contrast-Agents (GBCA) in Functional MR Urography (fMRU)
Brief Title: Gadolinium-Based-Contrast-Agents (GBCA) Enhancement During MR Urography
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Guerbet (Industry); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Aashim Bhatia, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: I002672
Record Dates: First submitted 2019-04-03; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Magnetic Resonance Imaging Contrast Agents
MeSH Terms: interventions — Gadolinium DTPA; gadoterate meglumine; gadobutrol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Dotarem Enhancement Group
  Interventions: Drug: Dotarem
- Gadovist Enhancement Group
  Interventions: Drug: Gadovist
- Magnevist Enhancement Group
  Interventions: Drug: Magnevist

INTERVENTIONS:
Drug: Magnevist — GBCA enhancement
  Groups: Magnevist Enhancement Group
Drug: Dotarem — GBCA enhancement
  Groups: Dotarem Enhancement Group
Drug: Gadovist — GBCA enhancement
  Groups: Gadovist Enhancement Group

SUMMARY:
Rationale: Dotarem provides superior enhancement characteristics compared to other GBCA in fMRU

Specific Aims: Compare enhancement characteristics of Dotarem to other GBCAs in the kidneys used in fMRU

Primary Objectives: Review functional analysis curves and data of fMRU studies and determine enhancement characteristics in the kidneys of the three GBCAs (Dotarem, Gadovist, Magnevist)

DETAILED DESCRIPTION:
A retrospective review will be performed of all functional MRI urography (fMRU) cases at two institutions (Children's Hospital of Philadelphia and Vanderbilt Children's Hospital). Over 1000 studies have been performed between the institutions and the normal studies will be selected based on radiology reports and reviewed to confirm they are normal. The fMRU is performed with Gadolinium based contrast agents (GBCAs), initially was performed with Magnevist, then switched to Gadavist, and most recently converted to Dotarem. The fMRU software for analysis of the functional data provides enhancement curves of the aorta and kidneys. fMRU enhancement curves are generated by drawing regions of interest in the aorta and renal parenchyma and calculating the average signal intensity over time. A comparison of the enhancement curves will be performed of the three GBCAs in the normal pediatric population. The enhancement curves will provide peak enhancement values within the aorta and kidneys (Time to peak = TTP) and allow comparison between the GBCAs. The enhancement intensity versus time will be evaluated for each GBCAs, providing an evaluation of how long renal parenchymal enhancement is maintained. Additional functional data will be reviewed such as calyceal transit time (CTT) and renal transit time (RTT).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric population which obtained MRI/fMRU study

Exclusion Criteria:

* Bilateral abnormal kidneys

Max Age: 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric population which obtained MRI/fMRU study
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 1990-07-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Dotarem TTP | 1 hour
  The enhancement curves will provide peak enhancement values within the aorta and kidneys (Time to peak = TTP) and allow comparison between the GBCAs.
Gadovist TTP | 1 hour
  The enhancement curves will provide peak enhancement values within the aorta and kidneys (Time to peak = TTP) and allow comparison between the GBCAs.
Magnevist TTP | 1 hour
  The enhancement curves will provide peak enhancement values within the aorta and kidneys (Time to peak = TTP) and allow comparison between the GBCAs.
Dotarem Time of Enhancement Intensity | 1 hour
  The enhancement intensity versus time will be evaluated for each GBCAs, providing an evaluation of how long renal parenchymal enhancement is maintained.
Gadovist Time of Enhancement Intensity Time of Enhancement Intensity for Gadovist | 1 hour
  The enhancement intensity versus time will be evaluated for each GBCAs, providing an evaluation of how long renal parenchymal enhancement is maintained.
Magnevist Time of Enhancement Intensity Time of Enhancement Intensity for Gadovist | 1 hour
  The enhancement intensity versus time will be evaluated for each GBCAs, providing an evaluation of how long renal parenchymal enhancement is maintained.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt Childeen's Hospital, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No